CLINICAL TRIAL: NCT05948917
Title: Mind-Body Skills Groups for Incarcerated Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Mind-Body Medicine (Other)
Collaborators: Herbert Simon Family Foundation (Unknown)
Responsible Party: Principal Investigator, Julie K. Staples, Research Director, The Center for Mind-Body Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMBMIndianaPrisons002
Record Dates: First submitted 2023-06-30; First posted 2023-07-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Resilience
Keywords: mind-body medicine; resilience; incarcerated; meditation; prisoners

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral: Mind-body Skills Groups (Experimental): 10 mind-body skills groups held once a week.
  Interventions: Behavioral: Mind-Body Skills Groups

INTERVENTIONS:
Behavioral: Mind-Body Skills Groups — The mind-body skills groups consist of supportive small group sessions with about 8-10 participants per group. Participants of these groups learn and practice mind-body techniques including: meditation, self-expression through drawings, autogenics and biofeedback, guided imagery, body awareness, and genograms.

SUMMARY:
The goal of this study is to learn about the effectiveness of a Mind-Body Skills Group program for incarcerated participants.The main questions is aims to answer are:

1. Do the mind-body skills groups increase resilience?
2. Do the mind-body skills groups decrease depression, anxiety and/or stress?
3. Do the mind-body skills groups increase participants' belief that they have improved coping skills?
4. Do the mind-body skills groups increase a sense of meaning in life?
5. Do the mind-body skills groups increase a sense of life purpose?
6. Do the mind-body skills groups increase self-esteem in women?
7. Do the mind-body skills groups decrease aggressive responses in men?

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for this study will be English-speaking incarcerated individuals at the Indiana Women's Prison and and at the Plainfield Correctional Facility.

Exclusion Criteria:

1. Having any of the following before the study is completed:

1. a sentence that will end,
2. a scheduled change in security level to a minimum-security prison or,
3. a scheduled work release;

Or 2. Having conduct problems and/or emotional or mental instability that prevents safe and effective participation in the mind-body medicine training program

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on resilience using the Connor-Davidson Resilience Scale (CD-RISC) after the 10-session mind-body skills groups and at 3 month follow-up. | Baseline, 11 weeks, and at 3 month follow-up
  The CD-RISC is a validated, self-report instrument assessing resilience over the last month. The CD-RISC consists of 25 questions that are rated on a 5-point scale with higher scores representing greater resilience.
  Change = After the 10 sessions score- Baseline score; Follow-up score - After the 10 sessions score; and Follow-up Score - Baseline score

SECONDARY OUTCOMES:
Change from Baseline on depression, anxiety, and stress using the Depression Anxiety and Stress Scale -21 (DASS-21) after the 10-session mind-body skills groups and at 3 month follow-up. | Baseline, 11 weeks, and at 3 month follow-up
  The DASS-21 is a validated, self-report instrument assessing the emotional states of depression, anxiety ans stress over the past week. The DASS-21 consists of 7 questions each for depression anxiety and stress are rated on a 4-point scale with higher scores representing higher levels of depression, anxiety, and stress.
  Change= After the 10 sessions scores- Baseline scores; Follow-up scores - After the 10 sessions scores; and Follow-up scores - Baseline scores
Change from Baseline on coping-self efficacy using the Coping Self-Efficacy (CSE) scale after the 10 session mind-body skills groups and at 3 month follow-up | Baseline, 11 weeks, and at 3 month follow-up
  The CSE Scale is a validated, self-report instrument assessing coping self-efficacy.
  The CSE scale consists of 26 questions that are rated on scale from 0 "cannot do at all" to 10 "certain can do". Higher scores represent greater levels of coping self-efficacy.
  Change = After the 10 sessions score- Baseline score; Follow-up score - After the 10 session score; and Follow-up score - Baseline score.
Change from Baseline on meaning in life using the Meaning in Life Questionnaire (MLQ) after the 10 session mind-body skills groups and at 3 month follow-up | Baseline, 11 weeks, and at 3 month follow-up
  The MLQ is a validated, self-report instrument assessing meaning in life. The MLQ consists of 10 questions that are rated on 7- point scale. There are 2 subscales: presence of meaning and search for meaning. Higher scores represent greater levels of these two components of meaning in life.
  Change = After the 10 sessions score- Baseline score; Follow-up score - After the 10 session score; and Follow-up score - Baseline score.
Change from Baseline on purpose in life using the the Life Engagement Test (LET) after the 10 session mind-body skills groups and at 3 month follow-up | Baseline, 11 weeks, and at 3 month follow-up
  The LET is a 6-item scale made up of items that are framed in half positive and half negative directions. These items are then rated using a 5-point scale that ranges from "1 = strongly disagree" to "5 = strongly agree".Higher scores represent greater levels of purpose in life.
  Change = After the 10 sessions score- Baseline score; Follow-up score - After the 10 session score; and Follow-up score - Baseline score.
Change from Baseline on self-esteem (females only) using the Rosenberg Self-Esteem Scale (RSE) after the 10 session mind-body skills groups and at 3 month follow-up | Baseline, 11 weeks, and at 3 month follow-up
  The RSE scale consists of 10 items scored on a 4-point scale with responses that range from "not at all like me" to "completely like me". Higher scores represent greater self-esteem.
  Change = After the 10 sessions score- Baseline score; Follow-up score - After the 10 session score; and Follow-up score - Baseline score.
Change from Baseline on aggression (males only) using the Aggression Questionnaire (AQ) after the 10 session mind-body skills groups and at 3 month follow-up. | Baseline, 11 weeks, and at 3 month follow-up
  Improvements in aggression will be measured using the Aggression Questionnaire (AQ) which is a revision of the Buss-Durkee Hostility Inventory that has been widely used to measure aggression.The AQ consists of 34 items scored on a 5-point Likert-type scale with responses ranging from "not at all like me" to "completely like me". The AQ has the following subscales: physical aggression, verbal aggression, anger, hostility, and indirect aggression. Higher scores represent greater aggression according to these components.
  Change = After the 10 sessions score- Baseline score; Follow-up score - After the 10 session score; and Follow-up score - Baseline score.

OTHER OUTCOMES:
How the Mind-Body Medicine Skills Groups have Affected the Participants by using Focus Group Interviews | 11 weeks
  Two focus groups with approximately with approximately 16-20 people each at each of the 2 prisons will be held. Focus group questions will cover topics such as how the mind-bdy skills groups have affected the participant in terms of relationships, how they view their future, and how they are going to used what they have learned.

CONTACTS AND LOCATIONS:
Overall Officials: Julie K Staples, PhD, Principal Investigator — The Center for Mind-Body Medicine
Locations (2):
- United States (2):
  - Plainfield Correctional Facility, Indianapolis, Indiana
  - Indiana Women's Prison, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No